CLINICAL TRIAL: NCT04874246
Title: Diluted VAsopressin During Robot-assisted Laparoscopic myomEctomy for dimiNishing Blood Loss According To the Dilution Concentration of Normal salINE: a Randomized Controlled Pilot Study
Brief Title: Comparison of Concentration of Vasopressin During Robot-assisted Laparoscopic Myomectomy
Acronym: VALENTINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: CHA University (Other)
Responsible Party: Principal Investigator, Hee Seung Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-107-1174
Record Dates: First submitted 2021-05-02; First posted 2021-05-05 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Uterine Leiomyoma
Keywords: Leiomyoma; Uterine fibroid; Uterine Myomectomy; Hemostasis; Vasopressin; Dilution
MeSH Terms: conditions — Myofibroma; Leiomyoma; Diabetes Insipidus | interventions — Vasopressins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diluted Vasopressin Group 1 (Active Comparator): During robot-assisted laparoscopic myomectomy, diluted vasopressin (a solution prepared by mixing 20 units of vasopressin with 50 ml of normal saline to make a total of 100 ml) was injected before uterine serosal incision.
  Interventions: Drug: Vasopressin
- Diluted Vasopressin Group 2 (Active Comparator): During robot-assisted laparoscopic myomectomy, diluted vasopressin (a solution prepared by mixing 20 units of vasopressin with 200 ml of normal saline to make a total of 100 m) was injected before uterine serosal incision.
  Interventions: Drug: Vasopressin
- Diluted Vasopressin Group 3 (Active Comparator): During robot-assisted laparoscopic myomectomy, diluted vasopressin (a solution prepared by mixing 20 units of vasopressin with 400 ml of normal saline to make a total of 100 m) was injected before uterine serosal incision.
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Vasopressin — During robot-assisted laparoscopic myomectomy, vasopressin diluted to different concentrations will be injected before uterine serosal incision.
  Other Names: Vasopressin 20U

SUMMARY:
The purpose of this study is to compare the effect of the concentration of vasopressin, which is used as a method for reducing blood loss in robot-assisted laparoscopic myomectomy.

DETAILED DESCRIPTION:
This study is to compare the effect of the concentration of vasopressin, which is used as a method for reducing blood loss in robot-assisted laparoscopic myomectomy. We would like to evaluate the feasibility and validity of this study for future Phase III randomized clinical trials through this preliminary randomized assignment study.

Uterine fibroids are the most common tumors in women, and uterine myomectomy, which is performed as a treatment for them, is basically a high risk of bleeding and blood transfusion. A common method to reduce intraoperative bleeding is to inject diluted vasopressin into the subserosal areas of the fibroids. However, no proper level of vasopressin dilution has been determined so far, so we want to determine an effective dilution concentration of vasopressin that can minimize side effects through this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age: 19-60 year-old women
* Plan of myomectomy for uterine leiomyomas
* Leiomyoma Subclassification System 2-7 (robot-assisted laparoscopic myomectomy is possible)
* American Society of Anesthesiologists Physical Status classification 1 or 2
* A person who understands the contents of the clinical trial, is cooperative with the trial, and is judged to be able to participate until the end of the study

Exclusion Criteria:

* Pregnancy or breastfeeding
* A single diameter of uterine leiomyoma is greater than 12 cm or more or multiple leiomyomas with more than five
* Suspicious disease of uterine malignancy
* Patient with has a history of pelvic surgery (cesarean section, myomectomy, etc.) and is expected to have severe pelvic adhesion
* A person who is hypersensitive or contraindicated to vasopressin
* A person who is hypersensitive or contraindicated to tranexamic acid
* Considered as inappropriate by the researcher's judgment

Ages: 19 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss (EBL) during operation | during operation
  The volume of blood loss will be estimated by using simple visual assessment technique referring to irrigation bottle

SECONDARY OUTCOMES:
Hemoglobin | Post-op 1 day
  Change of serum hemoglobin from baseline
Hematocrit | Post-op 1 day
  Change of serum hematocrit from baseline
Operation running time | during operation
  Time from anesthesia start to delivery of patient to recovery room
Transfusion | Post-op 2 days
  Whether patients are transfused during admission period Number of units transfused red blood cell
The amount of fluid injected during operation | during operation
  The amount of fluid injected during operation
Hospitalization period | Within post-op 1 week
  Days from admission day to discharge day

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, MD/PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park SJ, Lee JW, Hwang DW, Lee S, Yim GW, Song G, Lee EJ, Kim HS. Effect and Safety of Diluted Vasopressin Injection for Bleeding Control During Robot-assisted Laparoscopic Myomectomy in Reproductive Women With Uterine Fibroids: A Randomized Controlled Pilot Trial (VALENTINE Trial). In Vivo. 2024 Jan-Feb;38(1):431-436. doi: 10.21873/invivo.13456. PMID 38148064
- [Derived] Lee EJ, Park SJ, Kim Y, Lim H, Lee S, Yim GW, Song G, Kim HS. Effect and safety of diluted vasopressin injection on bleeding during robot-assisted laparoscopic myomectomy: a protocol for a randomised controlled pilot trial. BMJ Open. 2022 Sep 17;12(9):e056145. doi: 10.1136/bmjopen-2021-056145. PMID 36115677